CLINICAL TRIAL: NCT03099096
Title: An Open-label, Single Arm, Repeat Dose, Multi-centre Study to Evaluate the Use of an Autoinjector for the Subcutaneous Administration of Mepolizumab in Subjects With Severe Eosinophilic Asthma (Study 204959)
Brief Title: Study of Mepolizumab Autoinjector in Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204959; 2016-001832-36 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2018-06-29 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: SB240563; Mepolizumab; self-administration; eosinophilic asthma; autoinjector
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mepolizumab SC 100 mg/milliliter (mL) in autoinjector (Experimental): Three doses of mepolizumab liquid drug product in autoinjector will be self-administered by the subject/caregiver at 4-weekly intervals; 2 doses will be administered under observation in the clinic (at Week 0 and 8). One dose will be administered outside the clinic and without observation (within 24 hours after attending the clinic at Week 4).
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — It is a clear to opalescent, colorless to pale yellow sterile solution for SC injection, supplied in a single-use, prefilled syringe containing 100 mg/mL mepolizumab with sodium phosphate, citric acid, sucrose EDTA and polysorbate 80 within an autoinjector.

SUMMARY:
This study is aimed to assess the correct real-world use of an autoinjector for the repeat self-administration of mepolizumab SC, so to improve subject / physician convenience and to enable repeat dose self injection themselves or via caregivers. This Phase III study will be an open-label, single-arm, repeat-dose, multi-centre study of mepolizumab liquid drug product in autoinjector (100 milligrams [mg]) administered subcutaneously (SC) every 4 weeks (3 doses) in subjects with severe eosinophilic asthma. Subjects will receive 100 mg mepolizumab SC as a single injection that is self-administered in the thigh, abdomen or administered in the upper arm (caregiver only). Each subject will participate in the study for up to 18 weeks including pre-screening visit, a screening visit and a 12-week treatment period which concludes with end of study assessments (Visit 5) 4 weeks after the last dose of mepolizumab. Approximately 158 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 12 years of age inclusive, at the time of signing the informed consent. For those countries where local regulations permit enrolment of adults only, subject recruitment will be restricted to those who are >=18 years of age.
* Asthma: A physician diagnosis of asthma for >=2 years that meets the National Heart, Lung and Blood Institute guidelines or Global Initiative for Asthma guidelines.
* Mepolizumab treatment:

  a. Not receiving mepolizumab treatment at Visit 1. These subjects must also meet following inclusion criteria related to eosinophilic asthma, inhaled corticosteroid, controller medication and exacerbation history):
* Eosinophilic asthma: A high likelihood of eosinophilic asthma as per the required 'Continuation to Treatment'-criterion,
* Inhaled corticosteroid: A well-documented requirement for regular treatment with high dose inhaled corticosteroid (ICS) in the 12 months prior to Visit 1 with or without maintenance oral corticosteroids (OCS), for subjects >=18 years old, ICS dose must be >=880 micrograms (mcg)/day fluticasone propionate (FP) (ex-actuator) or equivalent daily, For ICS/long-acting-beta-2-agonist (LABA) combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion, for subjects >=12 to <=17 years old, ICS dose must be >=440 mcg/day FP (ex-actuator) or equivalent daily, for ICS/LABA combination preparations, the mid-strength approved maintenance dose in the local country will meet this ICS criterion. (Subjects will be permitted to be enrolled without continuous high dose ICS providing the subject was receiving continuous ICS and the Investigator attest that the subject should have been treated with high dose ICS to mitigate the risk of exacerbations, or the subject has financial or tolerance issues that prevent the use of high-dose ICS. Such subjects should be discussed with GSK Medical Monitor prior to enrolment)
* Controller medication: Current treatment with an additional controller medication, besides ICS, for at least 3 months or a documented failure in the past 12 months of an additional controller medication (e.g., LABA, leukotriene receptor antagonist [LTRA], or theophylline) for at least 3 successive months.
* Exacerbation history: Previously confirmed history of one or more exacerbations requiring treatment with systemic corticosteroid (CS) [intramuscular (IM), intravenous, or oral] in the 12 months prior to Visit 1, despite the use of high-dose ICS. For subjects receiving maintenance CS, the CS treatment for an exacerbation must have been a two-fold dose increase or greater.

or, b. Receiving 100 mg SC mepolizumab administered for the treatment of severe eosinophilic asthma every 4 weeks for at least 12 weeks prior to Visit 1.

* Body weight: A minimum body weight >=40 kilograms (kg) at Visit 1
* Gender: Male or female. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG)]test), planning to become pregnant during the time of study participation (and up to 16 weeks after the last dose), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: pre-menopausal females with documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or hysterectomy or documented bilateral oophorectomy, postmenopausal female, reproductive potential and agrees to follow highly effective methods for avoiding pregnancy in females of reproductive potential from 30 days prior to the first dose of study medication and until 16 weeks after the last dose of study medication and completion of the end of study/early withdrawal visit. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Informed consent: Capable of giving signed informed consent.

Exclusion Criteria:

* Concurrent respiratory disease: Presence of a known pre-existing, clinically important lung condition other than asthma. This includes current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Eosinophilic diseases: Subjects with other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, including churg-strauss syndrome, or eosinophilic esophagitis. Subjects with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 will also be excluded.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to screening. Subjects that had localized carcinoma of the skin which was resected for cure will not be excluded.
* Immunodeficiency: A known immunodeficiency (e.g. human immunodeficiency virus [HIV]), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Other concurrent medical conditions: Subjects who have known, pre-existing, clinically significant cardiovascular, endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Liver disease: Known, pre-existing, unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* ECG assessment: QT interval corrected for heart rate by either Fridericia's or Bazett's formula (QTc[F] or QTc[B]) >=450 milliseconds (msec) or QTc(F) or QTc(B) >=480 msec for subjects with bundle branch block at Visit 1.
* Xolair: Subjects who have received omalizumab within 130 days of Visit 1.
* Other monoclonal antibodies not including mepolizumab: Subjects who have received any monoclonal antibody to treat inflammatory disease within 5 half-lives of Visit 1.
* Investigational medications: Subjects who have received treatment with an investigational drug, other than mepolizumab within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to visit 1 (this also includes investigational formulations of marketed products) or experimental anti-inflammatory drugs (non biologicals) in the past 3 months.
* Chemotherapy: Subjects who have received chemotherapy within 12 months prior to Visit 1.
* Alcohol/substance abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.
* Hypersensitivity: Subjects with hypersensitivity to mepolizumab or to any of the excipients (sodium phosphate, citric acid, sucrose, ethylenediaminetetraacetic acid [EDTA], polysorbate 80).
* Adherence: Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- United States (16):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
- Australia (3):
  - GSK Investigational Site, Woodville South, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (4):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- Germany (5):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Russia (2):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Voronezh
- Sweden (2):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
- United Kingdom (5):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Background] Bernstein D, Pavord ID, Chapman KR, Follows R, Bentley JH, Pouliquen I, Bradford E. Usability of mepolizumab single-use prefilled autoinjector for patient self-administration. J Asthma. 2020 Sep;57(9):987-998. doi: 10.1080/02770903.2019.1630641. Epub 2019 Jun 28. PMID 31251090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with severe eosinophilic asthma, were enrolled at 16 sites in the United States of America, 6 sites in Germany, 5 sites in the United Kingdom, 4 sites in Canada, 3 sites in Australia, 2 sites in Russia and 2 sites in Sweden. The study duration lasted from 04 May 2017 to 30 November 2017.
Pre-assignment Details: Of the total 181 participants screened, 22 were screen failures and 159 were enrolled in this open-label, single arm, repeat dose study of mepolizumab and attempted to self-administer at least one dose of study treatment.
Groups:
- Mepolizumab Liquid Autoinjector: Participants (or their caregivers) self-administered, 100 milligram (mg) mepolizumab liquid drug product subcutaneously every 4 weeks (3 doses) as a single injection using autoinjector, in the thigh, abdomen or upper arm (caregiver only) for 12 weeks.
Period: Overall Study
Arm/Group | Mepolizumab Liquid Autoinjector
Started | 159
Completed | 157
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab Liquid Autoinjector
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (16.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 25
  Asian - Central/South Asian Heritage | 2
  Asian - East Asian Heritage | 1
  Asian - South East Asian Heritage | 3
  White - Arabic/North African Heritage | 1
  White - White/Caucasian/European Heritage | 126
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Self-administration of Their Observed Third Dose at Week 8 - Autoinjector With Standard Label + Pictogram
Description: Due to differences in the labelling requirements among regulatory authorities around the world, two different labelling approaches were included in this global study: labelling that includes a pictogram plus standard labelling elements, or a standard labelling without the pictogram. Participants (and/or their caregiver) attended three on treatment visits at Week 0, 4, 8, and End of Study Visit. Training on the study treatment, device handling and administration technique was provided by the investigator or qualified site staff at Week 0 and then first dose was self-administered under observation of investigator/site staff in clinic. Second dose self-administered unobserved, at home (Week 4) and third dose was self-administered under the observation of investigator/site staff in clinic (Week 8). All Subjects (Safety) Population included all enrolled participants attempting at least one self-administration of mepolizumab. Only participants with data available at Week 8 were analyzed.
Time Frame: Week 8
Population: All Subjects (Safety) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab Liquid Autoinjector
Number analyzed (Participants) | 103
Percentage of participants | 99

2. Primary Outcome: Percentage of Participants With Successful Self-administration of Their Observed Third Dose at Week 8 - Autoinjector With Standard Label Only
Description: Due to differences in the labeling requirements among regulatory authorities around the world, two different labeling approaches were included in this global study: labeling that includes a pictogram plus standard labeling elements, or a standard labeling without the pictogram. Participants (and/or their caregiver) attended three on treatment visits at Week 0, Week 4, Week 8, and the End of Study Visit. Training on the study treatment, device handling and administration techniques was provided by the investigator or qualified site staff at Week 0 and then first dose was self-administered under observation of investigator/site staff in clinic. Second dose self-administered unobserved, at home (Week 4) and third dose was self-administered under the observation of investigator/site staff in clinic (Week 8). Only participants with data available at Week 8 were analyzed.
Time Frame: Week 8
Population: All Subjects (Safety) Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Mepolizumab Liquid Autoinjector
Number analyzed (Participants) | 54
Percentage of Participants | 98

3. Secondary Outcome: Percentage of Participants With Successful Self-administration of Their Unobserved Dose at Week 4 - Autoinjector With Standard Label + Pictogram
Description: Due to differences in the labeling requirements among regulatory authorities around the world, two different labeling approaches were included in this global study: labeling that includes a pictogram plus standard labeling elements, or a standard labeling without the pictogram. Data for participants (and/or their caregiver) self-administering the second dose unobserved, at home (Week 4) using Autoinjector with Standard Label + Pictogram has been presented. Only participants with data available at Week 4 were analyzed.
Time Frame: Week 4
Population: All Subjects (Safety) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab Liquid Autoinjector
Number analyzed (Participants) | 103
Percentage of participants | 98

4. Secondary Outcome: Percentage of Participants With Successful Self-administration of Their Unobserved Dose at Week 4 - Autoinjector With Standard Label Only
Description: Due to differences in the labeling requirements among regulatory authorities around the world, two different labeling approaches were included in this global study: labeling that includes a pictogram plus standard labeling elements, or a standard labeling without the pictogram. Data for participants (and/or their caregiver) self-administering the second dose unobserved, at home (Week 4) using Autoinjector with Standard Label has been presented. Only participants with data available at Week 4 were analyzed.
Time Frame: Week 4
Population: All Subjects (Safety) Population
Measure: Number; unit: Percentage of participants
Arm/Group | Mepolizumab Liquid Autoinjector
Number analyzed (Participants) | 54
Percentage of participants | 96

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from start of Study Treatment (Week 0) until the End of Study/Early Withdrawal Visit (Week 12)
Description: On-treatment SAEs and non-serious AEs are reported for All Subjects (Safety) Population
Arm/Group | Mepolizumab Liquid Autoinjector
All-Cause Mortality (participants affected / at risk) | 0/159
Serious Adverse Events (participants affected / at risk) | 4/159
Other Adverse Events (participants affected / at risk) | 27/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab Liquid Autoinjector (N=159)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab Liquid Autoinjector (N=159)
Nasopharyngitis (Infections and infestations) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (5)
Headache (Nervous system disorders) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03099096/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03099096/SAP_001.pdf